CLINICAL TRIAL: NCT05818397
Title: Nurturing Compassionate Responding Towards Oneself and Others Through the Caregiver-child Relationship
Brief Title: Self-Compassion for Children and Caregivers
Acronym: SCCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Mind & Life Institute (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-0325; PEACEFP2022-9936264010 (Other Grant/Funding Number: Mind & Life Institute); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison); Protocol Version 11/27/2024 (Other: UW Madison)
Record Dates: First submitted 2023-04-03; First posted 2023-04-18 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Caregivers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Compassion Intervention - English speaking (Experimental)
  Interventions: Behavioral: Self-Compassion for Children and Caregivers (SCCC)
- Self-Compassion Intervention - Spanish speaking (Experimental)
  Interventions: Behavioral: Self-Compassion for Children and Caregivers (SCCC)

INTERVENTIONS:
Behavioral: Self-Compassion for Children and Caregivers (SCCC) — A standardized, manualized adaptation of the mindful self-compassion curriculum for adults, designed for online delivery. Dyads join a group video conference call along with other caregiver-child dyads and and up to two experienced SCCC facilitators. Sessions occur 1-hour per week for 6 weeks at a time convenient for the group.

SUMMARY:
The Self-Compassion for Children and Caregivers Study aims to understand if an online course designed to help kids and their caregivers learn self-compassion is feasible, enjoyable, and helpful for well-being and relationships in families from diverse backgrounds. Children ages 8-11 who have a caregiver willing to participate with them will:

* Attend 2 in-person study visits (about 1-1.5 hour each) that includes

  * A survey for caregiver and child
  * A brief computer puzzle challengetask while heart rate and sweat is recorded (child)
  * A brief discussion about how the challenge went
* Participate in a 6-session, online self-compassion course with other families (see back)
* Provide feedback about how the course went

DETAILED DESCRIPTION:
This pilot study examines the feasibility, acceptability, and preliminary outcomes of the Self-Compassion for Children and Caregivers (SCCC) program. Twenty-four children ages 8-11 and a primary caregiver will be recruited from a racially diverse school community to participate in 6 1-hour group intervention sessions over 6 weeks. Feasibility and acceptability data will guide program refinements; pre and post assessments will explore dimensional changes in anxiety/depression symptoms as well as potential physiological, relational/behavioral changes associated with SCCC participation.

ELIGIBILITY:
Inclusion Criteria - English speaking:

* Youth between the ages of 8 and 11 years old
* Youth are currently attending an elementary school in the Madison Metropolitan School District (MMSD).
* Accompanied by a willing and able caregiver (e.g., parent, grandparent, legal guardian)
* Access to an internet-enabled device
* Both parent and youth participants must be able to read/write in English
* Meet threshold (T greater than 59) for clinically significant anxiety and/or depression from either parent- or youth-report of symptoms

Inclusion Criteria - Spanish speaking:

* Youth between the ages of 8 and 11 years old
* Accompanied by an eligible caregiver participant
* Safe access to a computer or mobile device that can connect to the internet
* Visual acuity adequate to read text on a computer or mobile device
* Able to provide assent and complete surveys in Spanish

Exclusion Criteria - English speaking:

* Are unable to provide adequate informed consent and/or assent
* Parent or youth that is currently impaired by any medical condition that would prevent study participation
* Active self-reported psychotic disorder
* Current use of psychotropic medication is not exclusionary. However, certain medications that may impact physiology recordings may be excluded (e.g. those with direct impacts on the sympathetic nervous system). Exclusionary medications will be decided on a case-by-case basis, per discretion of the PI, a pediatric psychiatrist

Exclusion Criteria - Spanish speaking:

* Previous completion of a Mindfulness and Self-Compassion for children and Caregivers (MSC-CC) program

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Change in number of dyads in attendance each week | Week 1 to week 6
  Feasibility and acceptability will be measured using attendance records each week of the program
Reasons for study attrition | Up to week 6
  Feasibility and acceptability will be assessed through reasons provided by dyads for leaving the program
Fidelity to SCCC Curriculum | Through study completion, up to 2 years
  The SCCC Fidelity Checklist is a subjective checklist for evidence shown for an array of items covered during each session. No evidence, some evidence, and definite evidence are selected, with higher counts of definite evidence reflecting greater fidelity to the curriculum.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Herringa, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States